CLINICAL TRIAL: NCT00186342
Title: Allogeneic Sibling and Unrelated Donor Hematopoietic Cell Transplantation for Patients With Hematologic Malignancies Using Busulfan, Etoposide and Cyclophosphamide
Brief Title: Sibling and Unrelated Donor Hematopoietic Cell Transplant in Hematologic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robert Negrin, Professor of Lymphatic Research and Medicine, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT45; 75274; BMT45; NCT00186342
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Acute Disease; Myelodysplastic Syndromes; Leukemia, Myeloid, Chronic; Myeloproliferative Disorders; Blood and Marrow Transplant (BMT); Myelodysplastic Syndromes (MDS); Leukemia
MeSH Terms: conditions — Acute Disease; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myeloproliferative Disorders; Leukemia

ARMS (1):
- CIK cell (Experimental): The initial dose utilized will be 1x107 expanded cells/kg. The dose will be increased to 5x107 expanded cells/kg and 1x108 expanded cells/kg in successive escalations based on no significant infusional toxicity or GVHD.
  Interventions: Procedure: ablative allogeneic hematopoietic cell transplantation

INTERVENTIONS:
Procedure: ablative allogeneic hematopoietic cell transplantation

SUMMARY:
The purpose of this study is to determine the tolerability and efficacy in treating patients aged 51-60 with acute leukemia and in treating myelodysplastic syndromes (MDS) or myeloproliferative disorders (MPD).

DETAILED DESCRIPTION:
To learn whether a new preparative regimen to prepare patients for bone marrow transplantation is useful in patients above 50 years of age and whether it is useful in patients with myelodysplastic syndromes.

ELIGIBILITY:
Inclusion Criteria:1) Patients aged 51-60 with acute non-lymphocytic leukemia in first or subsequent remission and acute lymphocytic leukemia in first remission with high risk features which include elevated white blood cell count at presentation, cytogenetic abnormalities, extramedullary leukemia, ALL in greater than first remission and patients with chronic myelogenous leukemia at any stage who have a histocompatible sibling donor.

2) Patients with myelodysplastic syndrome including patients with refractory anemia with excess blasts or refractory anemia with excess blasts in transformation.

3) Patients with myeloproliferative disorders which give them poor long-term disease-free survival, such as myeloid metaplasia or myeloid fibrosis.

4) Patients with secondary myelodysplasia following cytotoxic chemotherapy. Exclusion Criteria:- Organ dysfunction

Ages: 51 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 1992-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
tolerability
efficacy of therapy

SECONDARY OUTCOMES:
compare efficacy of this treatment to historical controls

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Negrin, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States